CLINICAL TRIAL: NCT02559167
Title: Cannabidiol as a New Treatment for Cocaine Addiction
Brief Title: Cannabidiol and Cocaine Craving/Dependence
Acronym: CBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14.183
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-01

CONDITIONS: Substance Use Disorder; Cocaine Dependence; Withdrawal From Addictive Substance; Detoxification
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cannabidiol (Active Comparator): Participants will receive CBD 800 mg for 92 consecutive days starting on Day 2 of a 10-day inpatient detoxification period followed by 12 weeks of outpatient follow-up
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Participants will receive placebo for 92 consecutive days starting on Day 2 of a 10-day inpatient detoxification period followed by 12 weeks of outpatient follow-up
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — The investigators will carry out a double-blind, randomized, controlled trial comparing the effects of 92 days of 400 (only for the first 2 Days starting on the Day 2 of the study) or 800 mg CBD (subjects who report side effects with the 800mg dose will be administered the CBD 400 mg dose for the remainder of the trial) vs. placebo administration on cocaine craving and relapse in 110 cocaine-dependent subjects.
  Other Names: CBD

SUMMARY:
In this study, the investigators seek to evaluate the effects of cannabidiol (CBD) on cocaine craving and relapse. Cocaine addiction is characterized by compulsive substance use and repetitive urges to consume the drug even after a sustained period of abstinence. While substance use remains the most obvious direct outcome of addiction, there is a growing interest in other core symptoms of this disorder. Craving has become a subject of great interest as it is a reliable intermediate phenotype of cocaine relapse and a distressing symptom of addiction associated with suffering. Indeed, even after a period of abstinence, cocaine-dependent individuals remain vulnerable to stress and other craving-inducing stimuli, which, in turn, lead to intense physiological responses and various negative feelings such as anger and sadness. Real-time daily monitoring of craving and drug use has shown that craving predicts cocaine relapse among cocaine-dependent individuals. In sum, working toward improving the treatment of craving could not only help prevent relapse, but also reduce patient distress on emotional, cognitive, and physiological levels. In the past decades, significant scientific efforts have been deployed toward the development of innovative strategies to beat cocaine addiction, but with partial success thus far. Psychosocial approaches have been widely used to help cocaine-dependent patients achieve better outcomes after drug cessation, but literature indicates that these strategies alone are at times insufficient to induce significant behavioural changes or a reduction in rates of drug consumption. Unlike other types of addiction, such as opioid and alcohol, no pharmacological treatment has yet been found to be truly effective in relieving cocaine-cessation symptoms like craving and anxiety or to prevent relapse. CBD is a natural cannabinoid with a favourable tolerability profile and discrete neurobiological actions that are linked to neural circuits closely involved in addiction disorders. Addiction to cocaine is characterized by alternating phases of intoxication and short abstinence, followed by recurrent drug-craving episodes which result in distress and relapse. Our hypothesis is that CBD a cannabinoid known for its broad spectrum properties is an interesting pharmacological contender to decrease cocaine craving and treat cocaine addiction. Previous studies conducted in animals and humans confirm that CBD is a very safe and tolerable medication.

DETAILED DESCRIPTION:
The investigators will carry out a double-blind, randomized, parallel-group, placebo-controlled trial to assess the effects of 92 days of CBD 400 mg (for the first 2 days starting on Day 2 of the study) or 800 mg (subjects who report side effects with the 800mg dose will be administered the CBD 400 mg dose for the remainder of the trial) or placebo on cocaine craving and cocaine use among 110 cocaine-dependent individuals. Phase I of the trial will assess the effects of CBD or placebo administration on cocaine craving in the context of a 10-day inpatient medical detoxification period. Phase II of the trial will be a 12-week post-detoxification outpatient follow-up period.

ELIGIBILITY:
Inclusion criteria

* DSM-5 criteria for current cocaine use disorder (moderate or severe).
* Current cocaine use with last use during two weeks prior to admission to the study as confirmed by the Timeline Follow Back questionnaire.
* Age between 18 and 65 years old (inclusive).
* Women with diagnosed menopause (as confirmed by the study physician), under the age of 65, will be eligible for the study
* Subject consents to inpatient detoxification at the CHUM.
* Ability to give valid, informed consent.
* Ability to speak and read French or English.

Exclusion criteria

* Severe and/or unstable hepatic, neurologic (including diagnosis of seizures), cardiac (including arrhythmias) or renal disease), or any other severe or unstable medical condition that precludes safe participation in the study according to the study physician.
* Patients who are already immunocompromised (e.g., patients with human immunodeficiency virus-1 who do not meet the following criteria: undetectable HIV virus (using modern assay) and CD4 count >350 cells/uL in the last 6 months prior to enrolment, patients on antiretroviral therapy; or other infectious organisms), exhibit malignancy and/or have autoimmune syndromes.
* Hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal products.
* Severe psychiatric condition (history of schizophrenia, schizoaffective disorder or bipolar disorder); current acute psychosis, mania or severe suicidality based on the Mini International Neuropsychiatric Interview (MINI 7.0)).
* Pregnancy or breastfeeding.
* Inability (or unwillingness) of women of childbearing potential to use a medically acceptable form of contraception throughout study duration and for 3 months after dosing stops. A medically acceptable form of contraception is either: (1) contraceptive pill or intrauterine device or depot hormonal preparation (ring, injection, implant); and/or (2) a double barrier method of contraception such as diaphragm, sponge with spermicide and condom.
* Couples planning to conceive within the next 12 months.
* Men with history of fertility problems.
* Another current severe substance use disorder or any substance use disorder that would require pharmacological treatment according to the addiction specialist except nicotine (e.g. benzodiazepine or opiate for alcohol or opioid use disorder).
* Current treatment with medications that may interact with Cannabidiol (i.e., psychotropic medications such as benzodiazepines or anticonvulsants) or anticipation that the patient may need to initiate such treatment during the study.
* Any serious medical condition or psychiatric illness that precludes the subject from signing the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Drug-cue induced craving | Day 8
  A 10-point visual analog scale (VAS) used to measure craving responses in the context of cocaine cue-induced craving during the laboratory session on Day 8 of detoxification
Number of days to relapse | Day 10 to 92
  The number of days to relapse will be determined as the number of days between detoxification discharge (Day 10) and the day of first cocaine use as determined by the first positive urine test for cocaine (the day prior to urine testing will be entered as the day of relapse) or the first day of cocaine use self-reported by participants (the earliest of both measures)

SECONDARY OUTCOMES:
Stress-induced craving | Day 8
  A 10-point VAS used to measure craving responses in the context of stress-induced craving during the laboratory session on Day 8.
Cocaine use during the post-detoxification phase | Day 10 to 92
  The percentage of positive urine tests will be calculated - we will conservatively assign a 'positive' result to all visits for which the test result is not available for a given subject (including all visits after the subject's loss to follow-up and all scheduled 'intermediate' weekly visits to which the subject did not come or at which the test was not performed).

OTHER OUTCOMES:
Detailed cocaine craving | Day 1, Day 3, Day 5, Day 7, Day 9, Week 1, Week 3, Week 5, Week 7, Week 9, Week11
  Assessed using the Cocaine Craving Questionnaire: CCQ-Brief.
Subjective cocaine craving | Day 1, Day 3, Day 5, Day 7, Day 9, Week 1, Week 3, Week 5, Week 7, Week 9, Week11
  A 10-point VAS used to measure cocaine craving.
Cocaine withdrawal symptoms | Day 1, Day 3, Day 5, Day 7, Day 9, Week 4, Week 8, Week 12
  Assessed using the Cocaine Selective Severity Assessment: CSSA. The CSSA enquires about 18 symptoms commonly reported in the literature as being associated with early cocaine abstinence; items are rated on a scale of 0-7.
Anxiety | Day 2, Day 9, Week4, and Week 12
  Using the Beck Anxiety Inventory (BAI). 21-item self-report scale that measures the severity of anxiety in adults. The BAI total score is the sum of the ratings given by the examinee for the 21 symptoms. Each symptom is rated on a 4-point scale ranging from 0 to 3. The maximum score is 63 points.
Subjective anxiety | Day 1, Day 3, Day 5, Day 7, Day 9, Week 1, Week 3, Week 5, Week 7, Week 9, Week11
  A 10-point VAS used to measure anxiety.
Positive and negative affect | Day 1, Day 3, Day 5, Day 7, Day 9, Week 1, Week 3, Week 5, Week 7, Week 9, Week11
  Positive and Negative Affect Schedule: PANAS is a 10 positive and 10 negative affects rated on a scale from 1 to 5.
Blood pressure | Day 1 to 10, Week 4, Week 12
  Blood pressure during the laboratory session and daily during detoxification.
Heart rate | Day 1 to 10, Week 4, Week 12
  Heart rate during the laboratory session and daily during detoxification.
Self-report cocaine use during the post-detoxification phase | Day 10 to 92
  Total number of self-reported days of cocaine use using the Time Line Follow-Back (TLFB).
Sustained abstinence | Day 10 to 92
  Defined as three weeks without self-reported cocaine use (using the TLFB) or positive urine test
Addiction severity | Day 2 and Day 92
  Using the Addiction Severity Index: ASI-Lite questionnaire. The ASI-Lite is a semi structured interview tool to assess potential problem areas in substance-abusing patients: medical status, employment and support, drug use, alcohol use, legal status, family/social status, and psychiatric status.
Sleeping pills used during phase 1 (detoxification) | Day 1 to 10
  Doses of Benadryl or trazodone administered during detoxification.
Depressive symptoms | Day 2, Day 9, Week4 and Week 12
  Beck's Depression Inventory second edition: BDI-II. The BDI-II is a 21-item self-report instrument for measuring the severity of depression in adults.
Number of psychosocial intervention sessions (outpatient phase) | Day 10 to 92
  Number of attended group therapy sessions during the outpatient phase.
Compliance to CBD | Day 10 to 92
  Assessed by measuring CBD remaining in bottle weekly during post-detoxification visits and weekly journal entries by patient.
Completion rate | Day 10 to 92
  Assessed by determining if participants is still in the study at week 12.
Potential biological substrates of CBD's impact on cocaine craving and relapse - cortisol | Day 2, Day 8 and Week 4
  Assessed by measuring cortisol levels
Potential biological substrates of CBD's impact on cocaine craving and relapse - anandamide | Day 2, Day 8 and Week 4
  Assessed by measuring anandamide (AEA) levels
CBD plasma levels | Day 8, Day 9, Week 4 and Week 12
  CBD plasma levels.
Inflammatory markers - leukocytes | Day 2, Day 8, Week 4 and Week 12
  Assessed by evaluating modulation of the activation status of the immune cells (circulating leukocytes) in their sera at defined time points.
Inflammatory markers - inflammatory proteins | Day 2, Day 8, Week 4 and Week 12
  Assessed by evaluating modulation of the presence of inflammatory proteins in their sera at defined time points.
Cognition | Day 1, Day 7, Week 6
  Memory, attention, impulsivity and decision-making will be assessed using a CANTAB battery.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD,MS,FRCPC, Principal Investigator — Centre de Recherche du CHUM / Université de Montréal
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Hebert FO, Mongeau-Perusse V, Rizkallah E, Mahroug A, Bakouni H, Morissette F, Brissette S, Bruneau J, Dubreucq S, Jutras-Aswad D. Absence of Evidence for Sustained Effects of Daily Cannabidiol Administration on Anandamide Plasma Concentration in Individuals with Cocaine Use Disorder: Exploratory Findings from a Randomized Controlled Trial. Cannabis Cannabinoid Res. 2025 Apr;10(2):e341-e352. doi: 10.1089/can.2023.0273. Epub 2024 May 21. PMID 38770686
- [Derived] Mongeau-Perusse V, Rizkallah E, Morissette F, Brissette S, Bruneau J, Dubreucq S, Gazil G, Trepanier A, Jutras-Aswad D. Cannabidiol Effect on Anxiety Symptoms and Stress Response in Individuals With Cocaine Use Disorder: Exploratory Results From a Randomized Controlled Trial. J Addict Med. 2022 Sep-Oct 01;16(5):521-526. doi: 10.1097/ADM.0000000000000959. Epub 2022 Feb 8. PMID 35135986
- [Derived] Mongeau-Perusse V, Brissette S, Bruneau J, Conrod P, Dubreucq S, Gazil G, Stip E, Jutras-Aswad D. Cannabidiol as a treatment for craving and relapse in individuals with cocaine use disorder: a randomized placebo-controlled trial. Addiction. 2021 Sep;116(9):2431-2442. doi: 10.1111/add.15417. Epub 2021 Feb 9. PMID 33464660